CLINICAL TRIAL: NCT02814266
Title: Trakya University, Faculty of Medicine, Department of Anatomy, Edirne, Turkey
Brief Title: Difficult Intubation and Anthropometric Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, aliyilmaz, Principal Investigator, Assoc Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: TrakyaUniver
Record Dates: First submitted 2016-06-14; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Difficult Intubation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- difficult intubation (Other): Intubation difficulty score >5
  Interventions: Other: difficult intubation; Other: easy intubation
- Easy intubation (Other): Intubation difficulty score >5
  Interventions: Other: difficult intubation; Other: easy intubation

INTERVENTIONS:
Other: difficult intubation — Goniomastoid Distance: The distance between gonion and mastoid while the neck is fully extension and the mouth maximally open. Thyrogonial Distance: The distance between thyroidea and gonion while the neck is fully extension and the mouth maximally open.
Other: easy intubation — Goniomastoid Distance: The distance between gonion and mastoid while the neck is fully extension and the mouth maximally open. Thyrogonial Distance: The distance between thyroidea and gonion while the neck is fully extension and the mouth maximally open.

SUMMARY:
OBJECTIVE: This study aimed to determine the sensitivity and specificity of various anatomic measurements alone or in combination in predicting difficult intubation. The investigators hypothesized that goniomastoid distance, thyrogonial distance and tongue movements are sensitive and specific tests for predicting difficult intubation MATERIALS AND METHODS: The investigators included the data of 170 patients (85 difficult intubation and 85 easy intubation) who underwent an abdominal surgery under general anesthesia. Patients in difficult intubation (n=85) and easy intubation (n=85) groups were matched by age, BMI, and gender. Intubation difficulty scale (IDS) scores were recorded. Upward and downward maximal protrusions of tongue (UMPT and DMPT, respectively) were evaluated in all patients. Anthropometric measurements were measured.

DETAILED DESCRIPTION:
To define the tongue protrusion tests, anatomic landmarks and horizontal lines were used. The first horizontal line (lower target line) was passing through the midpoint of the distance between stomion to mentum (mandible height) and the second horizontal line (upper target line) was passing through the midpoint of the distance from subnasal to stomion (upper lip height). The horizontal lines were drawn with an erasable marker pen on the each patient's face. In the sitting position, patients were asked to make maximal tongue protrusion upward (UMPT) and downward (DMPT) in anatomical neutral position. The inability of the tip of the tongue to reach to the target line was scored "1" and ability of the tongue tip to reach or pass the target line was scored "2

ELIGIBILITY:
Inclusion Criteria:

* Undergoing abdominal surgery with general anesthesia
* Able to sit

Exclusion Criteria:

* Enable to sit,
* Patients had head or neck surgery,
* Patients with unstable cardiological and respiratory hemodynamic symptoms,
* Dental prosthesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
thyrogonial distance | 5 months
  thyrogonial distance in centimeter (cm)The distance between thyroidea and gonion while the neck is fully extension and the mouth maximally open.

SECONDARY OUTCOMES:
Goniomastoid distance | 5 months
  goniomastoid distance in centimeter(cm) The distance between gonion and mastoid while the neck is fully extension and the mouth maximally open.

IPD SHARING:
Plan to Share IPD: No